CLINICAL TRIAL: NCT01148927
Title: A Pilot Study to Evaluate the Quality of Life of Long Term Survivors of Adult Acute Lymphoblastic Leukemia
Brief Title: Quality of Life Study for Adult Patients With Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0619-CE
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Adult acute lymphoblastic leukemia patients

SUMMARY:
Acute lymphoblastic leukemia (ALL) accounts for about 20% of adult leukemias. Treatment results in adult ALL have lagged behind the improvements achieved in the pediatric population. A modified version of the Dana Farber Cancer Institute pediatric protocol is used to treat adult patients with ALL. The results seem to be superior to those reported with other adult protocols. However, there is limited data on the impact of such intensified approaches and resulting toxicities on the quality of life (QOL) of these survivors. Identifying important factors affecting the QOL may permit attempts at early interventions and may help to further modify the regimen and mitigate these adverse effects on QOL.

This study is evaluating the quality of life of long term survivors of adult ALL. It involves the patients filling out several questionnaires that are well-validated measures assessing various QOL issues of concern to these patients. The following questionnaires are used in this study:

* EORTC QLQ C30 to assess global health and major health domains
* Brief Pain Inventory (BPI)
* Personal Health Questionnaire (PHQ9) to assess psychosocial distress
* Functional Assessment of Cancer Therapy (FACT) Fatigue Questionnaire
* Peripheral Neuropathy Questionnaire

The data obtained from the questionnaires will be analyzed and the various domains of health will be quantified.

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed with adult ALL or T-lymphoblastic lymphoma
* Age >/= 18
* Have completed the two-year modified DFCI protocol at least three months earlier and are in continuous complete remission
* Understand English and are able to fill out questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Long-term survivors of adult acute lymphoblastic leukemia treated with modified Dana Farber Cancer Institute ALL protocol (91-01).
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2009-11; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the quality of life of the long-term survivors of adult acute lymphoblastic leukemia treated uniformly with the modified Dana Farber Cancer Institute ALL protocol (91-01) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Brandwein, MD, FRCPC, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada